CLINICAL TRIAL: NCT05324176
Title: Assessment of Diaphragm Thickness by Ultrasonography in Guillain Barre Syndrome and Myasthenia Gravis
Brief Title: Diaphragm Thickness by Ultrasonography in Neurological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MD.19.06.186.R1.R2
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Guillain-Barre Syndrome; Myasthenia Gravis
Keywords: diaphragm thickness
MeSH Terms: conditions — Guillain-Barre Syndrome; Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: Patients will be examined in the supine position. diaphragmatic thickness will is measured on both sides during a deep breath in inspiration and during expiration in the 3 groups: (1) Gillian-Barre syndrome; (2) Myasthenia Gravis; (3) control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gillian-Barre (Active Comparator): Patients will be examined in the supine position. diaphragmatic thickness will is measured on both sides during a deep breath in inspiration and during expiration.
  Interventions: Radiation: diaphragmatic ultrasound
- Myasthenia Gravis (Active Comparator): Patients will be examined in the supine position. diaphragmatic thickness will is measured on both sides during a deep breath in inspiration and during expiration.
  Interventions: Radiation: diaphragmatic ultrasound
- control (Active Comparator): Patients hospitalized with neurological disorders without affection of the respiratory system.
  Interventions: Radiation: diaphragmatic ultrasound

INTERVENTIONS:
Radiation: diaphragmatic ultrasound — diaphragmatic thickness will be measured on both sides during a deep breath in inspiration and during expiration.

SUMMARY:
participants will be allocated into three groups, acute neuropathy (Guillain Barre Syndrome) group, neuromuscular junction disorder(myasthenia gravis ) group, and control group(people with neurological disorders not affecting the respiratory system.Ultrasonography is done on the diaphragm. The index test (ultrasound imaging of the diaphragm) is used. A high-resolution portable ultrasound machine is used, with a 7- to 13-MHz linear array transducer. Patients will be examined in the supine position. diaphragmatic thickness will is measured on both sides during a deep breath in inspiration and during expiration. objectives: primary outcome: to compare diaphragm thickness between the three examined groups. Secondary outcome: correlation between clinical scores and reference US values of diaphragm

DETAILED DESCRIPTION:
after IRB (institutional research board ) approval, of the faculty of medicine, Mansoura University, Egypt, written informed consent from all participants will be taken. participants will be allocated into three groups, acute neuropathy (Guillain Barre Syndrome) group, neuromuscular junction disorder(myasthenia gravis ) group, and control group(people with neurological disorders not affecting the respiratory system. inclusion group: age more than 18, both sexes. exclusion criteria: cardiopulmonary disease, chest trauma, diaphragmatic injury, body mass index more than 30. Any participant who shows respiratory dysfunction on doing arterial blood gases and pulmonary function tests will not be enrolled in the study. methods: Ultrasonography is done on the diaphragm. The index test (ultrasound imaging of the diaphragm) is used. A high-resolution portable ultrasound machine is used, with a 7- to 13-MHz linear array transducer. Patients will be examined in the supine position. diaphragmatic thickness will is measured on both sides during a deep breath in inspiration and during expiration. objectives: primary outcome: to compare diaphragm thickness between the three examined groups. Secondary outcome: correlation between clinical scores and reference US values of diaphragm

ELIGIBILITY:
Inclusion Criteria:

* all adult patients admitted to the neurology department

Exclusion Criteria:

* cardiopulmonary diseases
* chest trauma
* diaphragmatic diseases
* Body Mass Index (BMI) > 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
diaphragm thickness | within 24 hours from hospital admission
  will be reported in (mm)

SECONDARY OUTCOMES:
Hughes clinical score | within 24 hours from hospital admission
  score of disability 1-5, "Hughes RA, Newsom-Davis JM, Perkin GD, Pierce JM.Controlled trial prednisolone in acute polyneuropathy.Lancet. 1978;2:750-3"

CONTACTS AND LOCATIONS:
Overall Officials: Aya M Zhran, Principal Investigator — Mansoura University Faculty of Medicine
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Not in US Or Canada, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Anonymous patients' data will be available with the PI or corresponding Author on reasonable request according to local IRB regulations
Time Frame: will be reported
Access Criteria: will be reported